CLINICAL TRIAL: NCT02948075
Title: Multicenter, Open-label Study of Safety and Efficacy of Quisinostat in Combination With Paclitaxel + Carboplatin Chemotherapy in Patients With Metastatic or Locally Advanced Epithelial Ovarian Cancer, Primarily Peritoneal or Fallopian Tube Carcinoma, Resistant to First Line Platinum and Paclitaxel Based Chemotherapy
Brief Title: Safety and Efficacy of Quisinostat, a Histone Deacetylase Inhibitor, in Combination With Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NewVac LLC (Industry)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-14-OvaII-1-QUI-2
Record Dates: First submitted 2016-10-24; First posted 2016-10-28 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2016-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — quisinostat; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Quisinostat 12 mg & Paclitaxel & Carboplatin (Experimental): One 3-weeks course includes 6 doses of Quisinostat 12 mg at Days 1, 3, 5, 7, 9 and 11 and Paclitaxel 175 mg/m2 and Carboplatin (mg/ml x min) x [GFR (ml/min) + 25] on Day 7 up to 6 cycles.
  Interventions: Drug: Quisinostat; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Quisinostat
  Other Names: JNJ-26481585
Drug: Paclitaxel
Drug: Carboplatin

SUMMARY:
This is a multicenter, open-label study of safety and efficacy of Quisinostat in combination with Paclitaxel + Carboplatin chemotherapy in patients with metastatic or locally advanced epithelial ovarian cancer, primarily peritoneal or fallopian tube carcinoma, resistant to first line platinum and Paclitaxel based chemotherapy.

The study will be carried out in 5-8 Russian and Belarusian sites. A maximum of 32 patients with metastatic or locally advanced epithelial ovarian cancer, primarily peritoneal or fallopian tube carcinoma, resistant to first line platinum and Paclitaxel based chemotherapy, will be enrolled in the study.

DETAILED DESCRIPTION:
The study will be consisted of screening period of 3 weeks before the beginning of Quisinostat administration, followed by the Investigational product treatment period of approximately 18 weeks (up to 6 cycles and 21 days for each cycle), a safety follow-up of 4 weeks after the last administration of the study therapy and post-treatment follow-up aimed at determination of progression-free survival, time to disease progression and overall survival rate in the study population.

An interim analysis will be performed after 10 patients are evaluated for efficacy. If 1 or less from 10 patients have an objective response (OR), the study will be stopped early for futility.

After screening and confirmation of inclusion/exclusion criteria, patients will be asked to come to the site to start taking Quisinostat.

All patients will receive Quisinostat in the dose of 12 mg on Day 1, 3, 5, 7, 9 and 11 of each treatment cycle. Administration of Paclitaxel and Carboplatin will be performed on Day 7 of each cycle. The cycles will be repeated once every 3 weeks (21 days).

In case of severe carboplatin hypersensitivity reaction, it is permitted to switch to Cisplatin (75mg/m2) as alternative to Carboplatin in the subsequent cycles.

Patients will receive up to 6 cycles of study therapy and then patients will continue to be followed-up for ORR, PFS, TTP, OS assessment in the study population.

The Post-treatment follow up will include:

* End of treatment visit will take place in case of treatment's completion within 6 cycles of study therapy.
* Early discontinuation visit will take place in case of the early study termination (before completion of 6 cycles) . The patients will be asked to make an Early discontinuation visit not later than in 4 weeks after administration of the last Investigational product dose.

After End of treatment or Early Discontinuation visit the patient will continue to be followed- for up to 1 year from the start of study treatment or until ICRR-determined progression (or death) (whichever is earlier). This will include tumor assessments every 6 weeks (±7 days).

Following disease progression, the Investigator will contact the patients or their relatives not less than once in 3 months in order to collect information concerning the patient's survival status and, cause of death. This will occur up to 1 year after initial start of treatment on this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Signed patient's information sheet and informed consent form to participate in the study.
2. Histological confirmed diagnosis of serous epithelial ovarian, primarily peritoneal or fallopian tube carcinoma.
3. Females aged ≥ 18 years.
4. Patients must have an ECOG status of 0 or 1.
5. Patients must have received only 1 prior line of platinum and Paclitaxel based chemotherapy.
6. Tumor progression observed not less than 1 month and no more than 6 months after completion of the planned number of cycles of first line platinum/Paclitaxel based chemotherapy (Carboplatin in the dose AUC5-6 or Cisplatin in the dose ≥ 75 mg/m2, in combination with paclitaxel for 6 q3-4 wk cycles) and indications for undergoing the second line chemotherapy.
7. The patients must have at least one measurable lesion according to RECIST 1.1 criteria.
8. Tissue block from archived material at diagnosis must be available and be submitted for predictive biomarker analysis.
9. Patient's ability to carry out visits and study procedures and to comply with the protocol.
10. Requirements for laboratory parameters determined below:

    Hematology: Absolute neutrophil count:

    Platelets:

    Hemoglobin: ≥ 1,500/mm3 (1.5 x 109 cells/L)
    * 100,000/mm3 (100 x 109 cells/L)
    * 9.0 g/dl Liver function: Total bilirubin: ≤ 1.5x upper limit of normal (ULN)

    Aspartate aminotransferase (AST) and alanine aminotransferase (ALT):

    Alkalinephosphatase:
    * 2.5x ULN, or ≤ 5.0 x ULN in the case of liver metastasis
    * 5.0 x ULN Renal function: Serum creatinine: ≤2 mg/dL Coagulation panel: Activated partial thromboplastin time (aPTT): ≤ 1.5 x ULN
11. The expected survival time not less than 6 months.
12. Women of childbearing potential (not sterile or in menopause less than 2 years) must be practicing an effective method of birth control during the whole period of the study and 6 months after the last administration of the investigational product. Effective methods include usage of a condom or diaphragm (barrier method) with spermicide.

Exclusion Criteria:

1. Patients previously treated with an HDAC inhibitor. Patients, who have been treated with Valproate for convulsions can be included, however only if the treatment has taken place > 30 days before the screening.
2. Have received treatment for ovarian cancer with any other prior chemotherapy than platinum (Carboplatin (AUC 5-6) or Cisplatin (≥ 75 mg/m2)) and paclitaxel (175-200 mg/m2) q3-4 wk for 6 cycles. Additional first line chemotherapy or prior treatment with additional investigational anticancer therapy is also an exclusion criterion.
3. Presence of specific toxicities of ≥ I grade, according to the NCI-CTCAE v.4.3, related to any prior anti-cancer therapy (excluding alopecia)
4. Patients with subsequent debulking operation (after first line chemotherapy) or radiotherapy due to the disease recurrence.
5. Patients who have undergone lower pelvis radiotherapy.
6. Patients with active or uncontrolled infection.
7. Patients with antibodies to human immunodeficiency virus (HIV), or hepatitis C virus (HCV), active hepatitis B virus (HBsAg).
8. History of other malignancies with the exception of basal cell carcinoma of the skin or cervical cancer in situ, that had undergone surgical removal or treatment within ≥ 5 years before the screening.
9. Patients with known cerebral metastases or clinical signs of cerebral metastases.
10. Have a history of severe hypersensitivity reaction to carboplatin, paclitaxel or agents within the histone deacetylase inhibitor group.
11. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess during the year prior to inclusion.
12. Clinically significant cardiovascular diseases including:

    * Myocardial infarction within 12 months before screening
    * Unstable angina within 12 months before screening
    * Congestive heart failure Class III or IV according to the New York Heart Association criteria (NYHA)
    * Clinically significant ventricular arrhythmia including ventricular tachycardia, ventricular fibrillation, history of cardiac arrest, atrioventricular block (Mobitz II or III), use of cardiostimulator
    * QTc interval > 470 ms (ECG) (calculated according to Fredericia formula), or a diagnosis of long QTc syndrome
    * Hypotension (systolic blood pressure < 86 mm Hg) or bradycardia with a heart rate of < 50 beats per minute (ECG) except when caused by medications (e.g. beta-blockers)
    * Uncontrolled arterial hypertension (systolic arterial pressure > 170 mm Hg or diastolic blood pressure > 105 mm Hg)
13. Pregnancy and lactation
14. Drug or alcohol abuse at the moment of screening or in the past which according to the opinion of the Investigator makes the patient unsuitable for participation in the study
15. Inability to read or write; inability to understand and comply with the procedures of the study protocol; failure to comply with the treatment, which, in opinion of the Investigator, may affect the results of the study or the patient's safety and prevent the patient from further participation in the study; any other associated medical or serious mental conditions that make the patient unsuitable for participation in the clinical study, limit the validity of informed consent or may affect the patient's ability to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Objective response rate | up to week 54
  assessment of the objective response rate ORR (complete response (CR) plus partial response (PR)) according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to week 54
Time to progression (TTP) | up to week 54
Overall survival (OS) | up to week 54
The percentage of patients in which the TTP1 on the first line chemotherapy with Carboplatin and Paclitaxel is shorter than TTP2 for the patients on second line chemotherapy with Carboplatin, Paclitaxel and Quisinostat | up to week 54
Determination of E-Cadherin, ERCC1 and BRCA1 expression as potential predictive biomarkers for Quisinostat induced sensitivity to chemotherapy | up to week 54
  the measurement will be conducted using tumor tissue samples
Incidence and severity of adverse events (AEs), including serious AEs (SAEs), graded according to the National Cancer Institute (NCI) CTCAE version 4.03 | up to week 54

CONTACTS AND LOCATIONS:
Overall Officials: Sergei A. Tjulandin, Prof., Principal Investigator — Russian Oncological Research Center n.a. N.N. Blokhin RAMS
Locations (6):
- Russia (6):
  - Federal State budget Scientific Agency "Russian Oncological Research Center n.a. N.N. Blokhin", Moscow
  - Medical Radiological Scientific Center n.a. A.F. Tsyb - branch of Federal State Budget Agency "Public Medical Scientific Radiology Center" of Ministry of Health of Russian Federation, Obninsk
  - State Budget Agency of Stavropol Territory Healthcare Pyatigorsk Oncologic Dispensary, Pyatigorsk
  - State Budget Agency of Healthcare "Leningradsky Regional Oncologic Dispensary", Saint Petersburg
  - State Budget Healthcare Agency "St-Petersburg clinical scientific-practical center of specialized types of medical care (oncology)", Saint Petersburg
  - St-Petersburg State Budget Agency of Healthcare "Municipal Clinical Oncological Dispensary", Saint Petersburg

IPD SHARING:
Plan to Share IPD: No